CLINICAL TRIAL: NCT04561492
Title: Exploratory Study Evaluating the Relevance of [68Ga]Ga -PentixaFor for Initial Staging and Therapeutic Evaluation of Symptomatic Multiple Myeloma Patients in First Line Treatment or in Relapse
Brief Title: Relevance of [68Ga]Ga -PentixaFor-PET for Initial Staging and Therapeutic Evaluation of Multiple Myeloma
Acronym: PentiMyelo
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC19_0289; 2024-516752-18-00 (EU CTIS Number)
Record Dates: First submitted 2020-09-03; First posted 2020-09-23 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga]Ga-PentixaFor (Experimental)
  Interventions: Drug: [68Ga]Ga-PentixaFor

INTERVENTIONS:
Drug: [68Ga]Ga-PentixaFor — Tomography by emission of positons (PET) with theradiopharmaceutic [68Ga]Ga-PentixaFor

SUMMARY:
The aim of our study is to confirm the relevance of PET using [68Ga]Ga -PentixaFor ligand, in comparison with FDG, for initial staging and therapeutic evaluation of symptomatic multiple myeloma patients in first line treatment or in relapse. The prognostic value of positive CXCR4 expression will also be assessed and [68Ga]Ga -PentixaFor/FDG discordances explored.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Symptomatic MM patients according to IMWG criteria (12) requiring first-line treatment
* Written and signed informed consent (obtained on the screening day at the latest and before any investigation)
* ECOG (Eastern Cooperative Oncology Group) < 2
* Patient affiliated to or beneficiary of the National Health Service

Exclusion Criteria:

* HIV positive, active Hepatitis B or C
* Childbearing or child breast feeding women
* Women or men without effective contraceptive barrier if needed
* eGFR < 50 ml/min by MDRD or CKDEPI
* Previous or concurrent second malignancy except for adequately treated basal cell carcinoma of the skin, curatively treated in situ carcinoma of the cervix, curatively treated solid cancer, with no evidence of disease for at least 2 years
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Known active infection
* Patient with uncontrolled insulin-dependent or non-insulin-dependent diabetes mellitus
* Patient under guardianship or trusteeship
* Patient under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2029-12-21 (Estimated); Study Completion 2030-05-21 (Estimated)

PRIMARY OUTCOMES:
To determine the sensitivity of [68Ga]Ga-PentixaFor-PET to detect Multiple Myeloma (MM) lesions [Bone marrow (BM) lesions and/or extra-medullary disease (EMD) ] at the time of initial diagnosis or at relapse. | 1 Month
  Sensitivity will be assessed by patient and lesion analysis by defining:
  * True positive (TP):
    * lesion positive with [68Ga]Ga-PentixaFor-PET and positive by FDG-PET
    * or lesion positive with [68Ga]Ga-PentixaFor-PET, negative on FDG-PET but confirmed by another CT scan/ MRI or histology, or confirmed by follow-up (until therapeutic evaluation).
  * False negative (FN): - lesion negative with [68Ga]Ga-PentixaFor-PET and positive by FDG-PET and confirmed by CT or MRI or histology, or confirmed by follow-up.

SECONDARY OUTCOMES:
To determine at the time of initial diagnosis or at relapse, the specificity, the positive predictive value (PPV) and negative predictive value (NPV) of [68Ga]Ga-PentixaFor-PET | 1 Month
  The specificity (PPV and NPV) of [68Ga]Ga-PentixaFor-PET at the time of initial diagnosis will be assessed by patient and lesion analysis using the same definitions of TP and FN as for the primary objective.
To determine at the time of initial diagnosis or at relapse, the prognostic impact of FDG PET and of [68Ga]Ga-PentixaFor-PET depending on the positivity, number and intensity of uptake detected by each imaging technique | 1 Month
  The prognostic impact of PET-FDG and [68Ga]Ga-PentixaFor-PET based on the number of lesions detected and their intensity of uptake by each imaging technique will be evaluated by assessing the impact of these data on the PFS and OS. PFS is defined as the time from the start of treatment to relapse or progression. OS is defined as the time from the start of first treatment to death.
To determine at the time of initial diagnosis or at relapse, the discrepancies rate between FDG PET and [68Ga]Ga-PentixaFor-PET | 1 Month
  Investigators will consider as discordant a lesion positive by FDG PET but negative by [68Ga]Ga-PentixaFor-PET and/or a lesion negative by FDG PET but positive by [68Ga]Ga-PentixaFor-PET
To determine at the time of initial diagnosis or at relapse, the factors associated with discrepancies between FDG PET and [68Ga]Ga-PentixaFor-PET | 1 Month
  Investigators will consider as discordant a lesion positive by FDG PET but negative by [68Ga]Ga-PentixaFor-PET and/or a lesion negative by FDG PET but positive by [68Ga]Ga-PentixaFor-PET
To determine at the initial diagnosis or relapse, the correlation between PET-FDG and [68Ga]Ga-PentixaFor-PET uptakes evaluated by SUV and the cytogenetic data evaluated on the myelogram (particularly the measurement of the expression of the gene coding | 1 Month
  68Ga]Ga -PentixaFor and FDG uptakes assessed by SUV and the quantitative expression of biological markers on myelogram (including expression of the gene coding for hexokinases).
To determine at the time of initial diagnosis or at relapse, the tolerance of [68Ga]Ga-PentixaFor-PET | 1 Month
  Tolerance of [68Ga]Ga-PentixaFor will be assessed by clinical monitoring of the patient for 1 hour after [68Ga]Ga-PentixaFor injection. Clinical data (heart rate, respiratory rate and blood pressure) will be collected prior [68Ga]Ga -PentixaFor injection before acquisition (at 60 min)
To determine at the time of initial diagnosis or at relapse, the tolerance of [68Ga]Ga-PentixaFor-PET | 1 Month
  Tolerance of [68Ga]Ga-PentixaFor will be assessed by clinical monitoring of the patientat the end of acquisition (at approximately 80 min).
To determine at the time of therapeutic evaluation the discrepancies rate between FDG PET and [68Ga]Ga-PentixaFor-PET and if available their link with histology. | 100 Day or 6 Month
  Investigators will consider as discordant a lesion positive by FDG PET but negative by [68Ga]Ga-PentixaFor-PET and/or a lesion negative by FDG PET but positive by [68Ga]Ga-PentixaFor-PET
To determine at the time of therapeutic evaluation the prognostic impact of FDG PET and [68Ga]Ga-PentixaFor-PET depending on the positivity, number and intensity of uptake detected by each imaging technique. | 100 Day and 6 Month
  The prognostic impact of [68Ga]Ga-PentixaFor-PET after therapy will be determined by evaluating the impact of a decrease uptake and/or a normalisation of images on PFS and OS.
To determine at the time of therapeutic evaluation the prognostic impact of FDG PET and [68Ga]Ga-PentixaFor-PET depending on the positivity, number and intensity of uptake detected by each imaging technique. | Every 6 months after the end of treatment
  The prognostic impact of [68Ga]Ga-PentixaFor-PET after therapy will be determined by evaluating the impact of a decrease uptake and/or a normalisation of images on PFS and OS.
To determine at the time of therapeutic evaluation the link between PET-FDG, [68Ga]Ga-PentixaFor-PET results and minimal residual disease evaluated by flow cytometry | 100 Day or 6 Month
  PET-FDG, [68Ga]Ga-PentixaFor-PET results (positive/negative) and minimal residual disease evaluated by flow cytometry (positive/negative).
To determine at the time of therapeutic evaluation the tolerance of [68Ga]Ga-PentixaFor-PET | 100 Day or 6 Month
  Tolerance of [68Ga]Ga-PentixaFor will be assessed by clinical monitoring of the patient for 1 hour after [68Ga]Ga -PentixaFor injection. Clinical data (heart rate, respiratory rate and blood pressure) will be collected prior [68Ga]Ga-PentixaFor injection before acquisition (at 60 min) and at the end of acquisition (at approximately 80 min).

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU Bordeaux, Bordeaux
  - CHU Lille, Lille
  - HCL, Lyon
  - Nantes UH, Nantes
  - APHP - Site Tenon, Paris

IPD SHARING:
Plan to Share IPD: Undecided